CLINICAL TRIAL: NCT01775592
Title: Monitoring the Efficacy of Dihydroartemisinin - Piperaquine in Patients With Uncomplicated Falciparum Malaria in Traleng Commune, Central Vietnam
Brief Title: Plasmodium Falciparum Artemisinin Resistance Vietnam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Malariology, Parasitology and Entomology, Vietnam (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMPE - ITM
Record Dates: First submitted 2013-01-11; First posted 2013-01-25 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Plasmodium Falciparum
Keywords: P.f resistance
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arterakin (Other): Number of DHA- PPQ (Arterakin™) tablets per day at 0hour, 8hours, 24hours, 48hours (according to age): 2 - 3 years:0.5, 0.5, 0.5, 0.5 3 - < 8 years: 1.0, 1.0, 1.0, 1.0 8 - < 15 years:1.5, 1.5, 1.5, 1.5
  ≥ 15 years:2.0, 2.0, 2.0, 2.0
  Interventions: Drug: Arterakin (DHA-PPQ)

INTERVENTIONS:
Drug: Arterakin (DHA-PPQ)

SUMMARY:
Resistance of Plasmodium falciparum toward Artemisinins, the most important drug for the successful treatment of malaria, has been confirmed in Cambodia. There are few reports from neighbouring countries about delayed parasite rates. The investigators therefore aim to assess parasite clearance in malaria patients in central Vietnam when treated according to national standard guidelines.

DETAILED DESCRIPTION:
General objective To evaluate the efficacy of DHA-PPQ in patients with uncomplicated falciparum malaria in a rural area of Central Vietnam, and to assess the in vitro susceptibility of P.falciparum isolates to DHA and PPQ.

Specific objectives

1. To measure the parasite clearance time in falciparum malaria patients treated with DHA-PPQ.
2. To determine the efficacy of DHA-PPQ at day 42 post-treatment.
3. To assess the in vitro susceptibility of P.falciparum isolates towards DHA and PPQ in Quang Nam Province.
4. To compare genetic profiles of P.falciparum isolates with delayed and those with normal clearance times in order to identify potential markers of resistance;

ELIGIBILITY:
Inclusion Criteria:

* Age: from 6 months of age;
* Fever (body temperature above 37.5C) or history of fever in the previous 24 hours;
* Mono-infection with P.falciparum with parasite density between 500-100,000/µl
* Written informed consent to participate to the trial. For patients aged less than 18 years, an informed consent will be obtained from a parent or a guardian.

Exclusion Criteria:

* Mixed malaria infection;
* Pregnancy or lactation (urine test for β human chorionic gonadotropin to be performed on any woman of child bearing age unless menstruating);
* Concomitant acute illness necessitating specific treatment (antibiotics);
* Underlying chronic severe illness (e.g. cardiac, renal, hepatic diseases, HIV/AIDS).
* Severe malnutrition;
* Danger signs:

  * not able to drink
  * incontrollable vomiting
  * recent history of convulsions (>1 in 24 hours)
  * unconscious state; neurological impairment
  * unable to sit or stand
* Signs of severe malaria:

  1. Cerebral malaria (unrousable coma)
  2. Severe anaemia (Htc< 15%)
  3. Renal failure (serum creatinine > 3 mg/dL)
  4. Pulmonary oedema;
  5. Hypoglycemia (<40mg/dL)
  6. Shock (systolic BP < 70 mmHg in adults, 50 in children)
  7. Spontaneous bleeding
  8. Repeat generalized convulsions
  9. Macroscopic haemoglobinuria
  10. Severe jaundice
* Persons who have received quinine, artemisinin or artemisinin derivatives within the last 7 days, 4-aminoquinolines within the last 14 days, pyrimethamine and/or sulfonamides within the last 28 days, or mefloquine within the last 56 days should be excluded from the in vitro testing

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Parasite clearance time | Day 2-5

SECONDARY OUTCOMES:
efficacy of DHA-PPQ at day 42 post-treatment in Traleng Quangnam, Vietnam | Day 42
  treatment failure or success at day 42
in vitro susceptibility of P.falciparum isolates towards DHA and PPQ in Quang Nam Province | Day 3-10
  MarkIII in vitro test

OTHER OUTCOMES:
genetic profiles of P.falciparum isolates with delayed and those with normal clearance times in order to identify potential markers of resistance | 1year
  genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Annette Erhart, MD, PhD, Principal Investigator — ITM
Locations (1):
- Health Centre Tra Leng, Tra Leng, Quang Nam, Vietnam

REFERENCES:
- [Derived] Thriemer K, Hong NV, Rosanas-Urgell A, Phuc BQ, Ha do M, Pockele E, Guetens P, Van NV, Duong TT, Amambua-Ngwa A, D'Alessandro U, Erhart A. Delayed parasite clearance after treatment with dihydroartemisinin-piperaquine in Plasmodium falciparum malaria patients in central Vietnam. Antimicrob Agents Chemother. 2014 Dec;58(12):7049-55. doi: 10.1128/AAC.02746-14. Epub 2014 Sep 15. PMID 25224002